CLINICAL TRIAL: NCT03627221
Title: The Effects of Combined Music Care With Sleep Management Network on Sleep Quality, Sleep Knowledge, and Sleep Hygiene in Nursing Students
Brief Title: Survey of Students' Sleep Related Outcomes and Sleep Management Network for Sleep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hui-Ling Lai, Professor, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB106-183-A
Record Dates: First submitted 2018-08-07; First posted 2018-08-13 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Sleep Quality
Keywords: social network; nursing students; sleep; music care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The intervention is social networking and music listening. The outcome variables are sleep quality, sleep knowledge, and sleep hygiene. The control variables are participants' demographic data.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A licensed sleep technician, blinded to group assignment, visually analyzed sleep polygraphs by applying standard procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music listening and social network (Experimental): The intervention group will receive music listening at sleep time and will be invited to join a social network for 12 weeks. But their sleep quality , sleep knowledge, sleep hygiene, daytime fatigue, and daytime sleepy will be collected for 12 months (at baseline, 3 month, 6 month, and the 12th month).
  Interventions: Behavioral: music listening and social network
- Control group (No Intervention): The control group will not receive music listening at sleep time and will not be invited to join a social network for 12 weeks. But their sleep quality, sleep knowledge, sleep hygiene, daytime fatigue, and daytime sleepy will be collected for 12 months (at baseline, 3 month, 6 month, and the 12th month).

INTERVENTIONS:
Behavioral: music listening and social network — The 12-week combination of music care and social network program consists of three parts: sleep related variables assessment and monitoring, sleep management education and outcome evaluation. Participants in the intervention group will receive weekly online (social network) education and music listening interventions for 12 weeks provided by the PI.
  Arms: music listening and social network

SUMMARY:
Several factors may cause sleep disturbance among nursing students. Sleep and its several influencing factors are both continuous dynamic process. However, research related to sleep and related issue in nursing students in a longitudinal manner is limited worldwide. Thus, the investigators intend to conduct a 3-year research divided into three phases to explore the issue. The first phase will adopt longitudinal panel study design. Nursing students from two schools will be invited to participate in the first year study, which will be about 800 people. The second phase is to classify music appreciated by the students into different music quadrants that may be effective and can be used at the third phase. The third phase is designed to explore the longitudinal effects of a 3-month social network combined with music care program on sleep quality, sleep knowledge, sleep hygiene and daytime sleepiness and fatigue. Students will be randomized into 2 groups: intervention and control groups. Participants in the intervention group will receive a 12-week intervention program. The control group will be no intervention. Growth curve modeling will be employed in this study for longitudinal analyses to identify the sleep predicted by the students' characteristics. This study will enable us to advance knowledge and research about nursing students' longitudinal patterns of sleep and the longitudinal effects of the intervention program on their sleep.

DETAILED DESCRIPTION:
Background: Poor sleep quality affect students' learning achievement. Several factors may cause sleep disturbance among nursing students. Sleep and its several influencing factors are both continuous dynamic process. However, changes in students' sleep patterns and related characteristics over time remain unclear. Therefore, understanding the issue and examining an effective program is important to ameliorate sleep and improve learning. Integrated care program has proved to be a nursing students' health promotion intervention. However, research related to sleep and related issue in nursing students in a longitudinal manner is limited worldwide. Thus, the investigators intend to conduct a 3-year research divided into three phases to explore the issue. Objectives: The first phase will adopt longitudinal panel study design. Nursing students from two schools will be invited to participate in the first year study, which will be about 800 people.The data will be obtained from 4 waves (the interval of each wave will be 2 months) of the longitudinal survey of sleep quality of the nursing students and how the students' characteristics influence sleep. Distinct patterns of sleep over time will help to identify what characteristics of students to target for the researchers and to make evidence-based intervention for them. The second phase is to classify music appreciated by the students that may be effective and can be used at the third phase. The third phase is designed to explore the longitudinal effects of a 3-month social network combined with music care program on sleep quality, sleep knowledge, sleep hygiene and daytime sleepiness and fatigue. 100 students will be randomized into 2 groups: intervention and control groups. Participants in the intervention group will receive a 12-week intervention program. The control group will be no intervention. Data will be collected from both groups at pretests, and at different time points depending on variables after intervention completed. Statistical analysis: Growth curve modeling will be employed in this study for longitudinal analyses to identify the trajectory of sleep predicted by the students' characteristics. Descriptive analyses will be conducted using SPSS 18. Anticipated results and implications: This study will enable us to advance knowledge and research about nursing students' longitudinal patterns of sleep and the longitudinal effects of the intervention program on their sleep. If the longitudinal effects of the intervention program on their sleep are confirmed, the findings will provide evidence for educators and policy makers using evidence-based intervention to ameliorate sleep in nursing students.

ELIGIBILITY:
Inclusion Criteria:

poor sleep quality (PSQI > 5)

Exclusion Criteria:

* pregnancy
* currently receiving stress management programs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
sleep quality | 18 months (intervention will last for 12 weeks)
  participants' subjective sleep quality will be measured by using the Pittsburgh Sleep Quality Index (PSQI). The PSQI has 19 items, most with a 4-point, Likert-type response scale. The total score of the 19 items is ranged between 0-21. The higher scores (greater than 5) indicate the participants have poorer sleep quality.

SECONDARY OUTCOMES:
sleep knowledge | 18 months (intervention will last for 12 weeks)
  The investigators developed questionnaire of sleep knowledge is a 10-15 questions regarding sleep-related knowledge. Each item oﬀered three response options: yes, no, or unsure. One point was assigned for a correct response, and zero was assigned for incorrect or "unsure" responses. The maximum score was 10-15 points. The total score was treated as a global indicator of the levels of the participants' sleep knowledge. A higher score indicated that they were more knowledgeable about sleep.
sleep hygiene | 18 months (intervention will last for 12 weeks)
  Sleep Hygiene Index (SHI) will be used to measure participants' practice of sleep hygiene behaviors. The SHI is a 13-item self-report rated on a five-point scale ranging from 0 (never) to 4 (always). Total scores range from 0 to 52, with a higher score representing poorer sleep hygiene.
daytime fatigue | 18 months (intervention will last for 12 weeks)
  Daytime fatigue will be measured by using a 7-item scale, Flinders Fatigue Scale.
  Six items are presented in Likert format, with responses ranging from 0 (not at all) to 4 (extremely). Item 5 measures the time of day when fatigue is experienced and uses a multiple-item checklist. Total fatigue is calculated as the sum of all individual items. Total fatigue scores range from 0 to 31, with higher scores indicating greater fatigue.
daytime sleepiness | 18 months (intervention will last for 12 weeks)
  The Epworth Sleepiness Scale (ESS), a self-report 8-item questionnaire will be used to measure daytime sleepiness. The ESS is a four-point rating scale. Response categories range from "0 = would never doze," "1 = slight chance of dozing," "2 = moderate chance of dozing," "3 = high chance of dozing." Ratings are added over the eight items for a total score. The range of possible scores is from 0 to 24 points.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Lai, PhD, Principal Investigator — Tzu Chi University
Locations (1):
- Tzu Chi University, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No